CLINICAL TRIAL: NCT02570139
Title: Multi-Center, Randomized Trial Comparing the Efficacy of 3M™ Cavilon™ Advanced Barrier Film for the Treatment of Incontinence-associated Dermatitis to a Commercially Available Moisture Barrier
Brief Title: Clinical Study to Assess a New Barrier Film's Ability to Provide Skin Protection Against Incontinence & Allow Healing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment, short stay; lacked statistically powered evaluation for efficacy.
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EM-05-012990
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Incontinence Associated Dermatitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cavilon Advanced Skin Protectant (Experimental): Product applicator contains liquid barrier applied on buttocks/thighs with it drying rapidly to durable barrier film. It's applied 3x/per week.
  Interventions: Device: Cavilon Advanced Skin Protectant
- ConvaTec Sensi-Care Protective Barrier (Active Comparator): Marketed product applied following manufacturer's recommendation. The product is 15% zinc oxide with petrolatum.
  Interventions: Device: ConvaTec Sensi-Care Protective Barrier

INTERVENTIONS:
Device: Cavilon Advanced Skin Protectant — The liquid barrier film flows from the applicator and dries quickly on the skin. It is durable for 72-96 hours under conditions of incontinence.
  Arms: Cavilon Advanced Skin Protectant
Device: ConvaTec Sensi-Care Protective Barrier — Sensi-Care is commercial paste product applied to protect denuded and weeping skin from incontinence.
  Arms: ConvaTec Sensi-Care Protective Barrier

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of the investigational product (3M™ Cavilon™ Advanced High Endurance Skin Protectant) for the treatment of incontinence associated dermatitis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluated the product performance of a new skin protectant formulated to protect damaged and denuded skin even in the presence of exposure to the most potentially damaging body fluids, such as liquid stool and gastric fluid. The product is expected to intimately adhere to damaged and denuded skin and provide better protection from further damage than commonly used products such as moisture barrier pastes, thereby making it easier for nursing staff to cleanse the skin after incontinence episodes, thus saving time and also materials.

The denuded sites on buttocks/thighs will be scored for skin loss and degree of redness. Over the course of time, with the skin protected, it should re-epithelizes. The skin improvement will be scored and the change in baseline over time monitored.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be enrolled into this study if the answers to all these questions are yes.

1. Is the subject a full-term newborn (36 weeks or greater gestational age) or older?
2. Is the subject in a facility providing nursing care 24 hours per day?
3. Does the subject have severe Category 2 Incontinence-Associated Dermatitis (IAD) -red with skin breakdown (i.e. skin erosion and denudation or denudation of skin alone)?
4. Is the subject willing to have photos taken of their skin exposed to incontinence and permit use of photographs in potential publication?
5. Is the subject willing to release rights to 3M for the use of the photos?
6. Is there a reasonable expectation that the subject will remain in a facility for at least 7 days following enrollment in the study?
7. Has the subject, or their legally authorized representative, signed an Institutional Review Board-approved informed consent/assent document and authorized the use and disclosure of protected health information?

Exclusion Criteria:

* Subjects are excluded from participation in this study if any of the answers to these following questions is yes.

  1. If female, is the subject pregnant or breast feeding or has she given birth within the 3 weeks preceding the screening visit?
  2. Does the subject have a known allergy to acrylates or cyanoacrylates?
  3. Does the subject have a Stage III, IV, unstageable, suspected deep tissue injury pressure ulcer in the area where the skin is affected by incontinence?
  4. Does the subject have a preexisting skin disease on the areas affected by incontinence that may make skin assessments for this study difficult?
  5. Does the skin area affected by incontinence require treatment with a concomitant medication or product?
  6. Does the subject have an active genital herpes infection?
  7. Has the subject received antifungal powders in the area affected with IAD within 24 hours prior to enrollment?
  8. Has the subject received cyanoacrylate based skin protectant (such as Marathon) within 72 hours prior to enrollment?
  9. Is the facility unwilling to discontinue use for this subject of Dimethicone-containing wipes on the area where the skin protectant product will be applied?
  10. Is the facility unwilling to discontinue use for this subject of Chlorhexidine Gluconate wipes on the area where the skin protectant product will be applied?
  11. Does the subject have any medical condition that in the opinion of the investigator should exclude him/her from participating in the study?
  12. Has the subject been enrolled in any investigational study where product was applied to proposed study sites within 30 days of the screening visit?

Min Age: 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pat Parks, MD, Study Director — 3M
Locations (10):
- United States (10):
  - Children's Hospitals and Clinic, Minneapolis, Minnesota
  - Children's Hospital and Clinics, Saint Paul, Minnesota
  - Good Samaritan, Kearney, Nebraska
  - St. Elizabeth, Lincoln, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - Lennox Hill, New York, New York
  - St. John, Tulsa, Oklahoma
  - Roper St. Francis, Charleston, South Carolina
  - Baylor Plano, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cavilon Advanced Skin Protectant | ConvaTec Sensi-Care Protective Barrier
Started | 24 (24 subjects were treated w/ Cavilon Advanced Skin Protectant. Study terminated due to low enrollment) | 21 (21 subjects treated with SensiCare Protective Barrier)
Completed | 24 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patient with IAD, Category 2 (denuded skin)
Groups:
- Cavilon Advanced Skin Protectant: Product applicator contains liquid barrier applied on buttocks/thighs with it drying rapidly to durable barrier film. It's applied 3x/per week.
  Cavilon Advanced Skin Protectant: The liquid barrier film flows from the applicator and dries quickly on the skin.
- Total: Total of all reporting groups
Arm/Group | Cavilon Advanced Skin Protectant | ConvaTec Sensi-Care Protective Barrier | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Customized [Mean (Standard Deviation); unit: years or weeks] — adults are measured in years Population: The age distribution is between years for adults
  years or weeks
    Years: number analyzed (Participants) | 21 | 18 | 39
    Years | 67.1 (19.33) | 62.1 (19.97) | 64.8 (19.54)
Age, Customized [Mean (Standard Deviation); unit: Weeks] — Weeks of pediatrics Population: the discrepancy in overall number of baseline patients is due to revised age of the pediatric patients (in weeks) vs adult population (years). The total number of participants is unchanged.
  Weeks
    Weeks: number analyzed (Participants) | 3 | 3 | 6
    Weeks | 11.3 (7.37) | 20.3 (4.51) | 15.8 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 14 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 20 | 21 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 17 | 18 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 21 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to End of Study in Incontinence Associated Dermatitis (IAD) Scores
Description: Primary endpoint was percent decrease in Incontinence Associated Dermatitis (IAD) score from baseline to end of subject's participation. A negative value indicates increased IAD score; a positive value indicates decreased IAD score. IAD scores were calculated for 6 anatomical zones for color, presence of lesions, and skin loss using 3M's Skin Condition Assessment Tool. Skin condition assessed for 1) epidermal loss depth & area involved; 2) skin color intact skin & % area if not normal color. Intensity scored based on % area involved. Epidermal loss intensity rating scores ranged from 0 (none) - 4 (76-100%) partial (skin open, not weeping) or complete (skin open & weeping). Color of intact skin rating scores ranged from 0 (skin color normal) - 4 (76-100%) skin color pink or red. Scores for each of the 6 body zones were combined to obtain a single IAD score for each subject. IAD scores ranged from 0 (best) - 720 (worst).
Time Frame: up to 21 days depending on length of hospitalization
Population: Analysis was done using the intent-to-treat (ITT) population, using all subjects who had at least one dose of their assigned product.
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Cavilon Advanced Skin Protectant | ConvaTec Sensi-Care Protective Barrier
Number analyzed (Participants) | 24 | 21
percentage change | 11.0 (13.2) | 34.3 (14.1)

2. Secondary Outcome: Re-epithelialization to a Category 1 or Lower
Description: Looking for healing of denuded skin to re-epithelialized skin.
Time Frame: Up to 21 days depending on length of hospitalization
Population: Review and analysis of healing of denuded skin to re-epithelialization.
Measure: Count of Participants; unit: Participants
Arm/Group | Cavilon Advanced Skin Protectant | ConvaTec Sensi-Care Protective Barrier
Number analyzed (Participants) | 25 | 21
Participants | 6 | 5

3. Secondary Outcome: Pain Scores During Incontinence Management
Description: Pain scores during incontinence management were measured on a 0-10 scale, and analyzed only for subjects from the intent-to-treat dataset who could report pain. Adult pain was measured on 0-10 Wong-Baker FACES® Pain Scale Visual Analog to see if there is pain reduction (0 - no pain; 10 - worst pain). Pain in pediatric patients was measured with the 0-10 FLACC (Face, Legs, Activity, Cry, Consolability Behavioral) Tool. FLACC tool scores pain based on 5 categories, each scored on 0-2 scale and a total score calculated from the sum of the 5 categories for a total possible 0 (no pain) - 10 (worst pain) score. Data from the 2 scales were combined for analysis. Reduction in pain scores collected during product application were reported and least squares means adjusted for baseline pain score as a covariate were calculated. Negative value indicates reduction in pain score; positive value indicates increased pain score.
Time Frame: Up to 21 days depending on length of hospitalization
Population: The patient population analyzed were those who could report pain
Measure: Least Squares Mean (Standard Error); unit: Change in Score on 0-10 Scale
Arm/Group | Cavilon Advanced Skin Protectant | ConvaTec Sensi-Care Protective Barrier
Number analyzed (Participants) | 13 | 11
Change in Score on 0-10 Scale | -0.7 (0.8) | 0.3 (1.0)

4. Secondary Outcome: Prevention of IAD.
Description: Number of subjects with areas of buttock and thighs that were free of IAD at baseline and remained free of damage with ongoing incontinence through 5 days of treatment.
Time Frame: Measured at study day 5
Population: This is the population who went thru 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cavilon Advanced Skin Protectant | ConvaTec Sensi-Care Protective Barrier
Number analyzed (Participants) | 9 | 7
Participants | 8 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data was captured for 1 year, 9 months.
Arm/Group | Cavilon Advanced Skin Protectant | ConvaTec Sensi-Care Protective Barrier
All-Cause Mortality (participants affected / at risk) | 1/24 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/24 | 3/21
Other Adverse Events (participants affected / at risk) | 2/24 | 3/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cavilon Advanced Skin Protectant (N=24) | ConvaTec Sensi-Care Protective Barrier (N=21)
Gi Bleed (Gastrointestinal disorders) | 0 | 1
Hypotension (Cardiac disorders) | 0 | 1
Non-occlusive thombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cavilon Advanced Skin Protectant (N=24) | ConvaTec Sensi-Care Protective Barrier (N=21)
fungal infection (Skin and subcutaneous tissue disorders) | 2 | 2
Eczematous eruptions on back/arms (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT02570139/Prot_SAP_000.pdf